CLINICAL TRIAL: NCT03975959
Title: Prospective and Retrospective Memory Perception Assessment in Central/Non-central Nervous System Cancers
Brief Title: Memory Perception Assessment in Central/Non-central Nervous System Cancers
Acronym: PROMESSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: PROICM 2018-07 BPR
Record Dates: First submitted 2019-05-27; First posted 2019-06-05 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Glioblastoma; Glioma; Breast Cancer; Healthy
Keywords: PROMESSE; PROSPECTIVE MEMORY; RETROSPECTIVE MEMORY
MeSH Terms: conditions — Glioblastoma; Glioma; Breast Neoplasms | interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Intervention Model Description: The protocol administration will take about 20 minutes. It will be conducted by an experienced clinical neuropsychologist or clinical oncologist in each center during standard care. According to the results on the questionnaires and test, patients will be addressed and managed by a neuropsychologist, a clinical psychologist, psychiatrist or a speech therapist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GLIOBLASTOMA (Other): One visit with collection :
  demographical data clinical data QMRP questionnaire HADS questionnaire MFI questionnaire MoCA test FAB test
  Interventions: Other: QMRP questionnaire
- glioma (Other): One visit with collection :
  demographical data clinical data QMRP questionnaire HADS questionnaire MFI questionnaire MoCA test FAB test
  Interventions: Other: QMRP questionnaire
- breast cancer (Other): One visit with collection :
  demographical data clinical data QMRP questionnaire HADS questionnaire MFI questionnaire MoCA test FAB test
  Interventions: Other: QMRP questionnaire
- healthy (Other): One visit with collection :
  demographical data clinical data QMRP questionnaire HADS questionnaire MFI questionnaire MoCA test FAB test
  Interventions: Other: QMRP questionnaire

INTERVENTIONS:
Other: QMRP questionnaire — a single consultation for test and questionnaires for a duration of 20 minutes
  Other Names: HADS questionnaire; MFI questionnaire; MOCA test; FAB test

SUMMARY:
Prospective memory (PM) is the ability to implement intended actions in the future. It allows maintaining and retrieving future plans, goals, and activities (i.e., remember to remember). PM is associated with most everyday memory problems . PM is crucial to correctly respond to all the social, occupational and working demands of everyday life, to perform many deferred health-related actions and is involved in therapeutic adherence .

Indeed, PM errors are an important part of the aging memory complaints. The prevalence of self-reported PM failures is also significant among young adults, compared with self-reported retrospective memory (RM) failures .Yet, PM errors are major sources of frustration and embarrassment .

In oncology, recently investigated the self-reported memory complaints in a 80 case-healthy-control study breast patients . Subjective memory complaints were assessed using the Prospective and Retrospective Memory Questionnaire . Results from the Paquet et al. study show that all participants (i.e., both patients and matched-controls) reported more PM than RM failures in daily-life (p<.001). Breast cancer patients reported more RM and PM failures than controls. However, this group effect was no longer statistically significant when controlling for depression and fatigue.

These findings are consistent with the view that memory complaints are closely associated with depression and cancer-related fatigue, and more generally with psychopathological variables .As underlined by Paquet et al. subjective memory complaints should be investigated because they refer to some aspects of the cancer experience that could potentially be linked to quality of life. Thus, it is important to explore psychopathological basis such as depression, anxiety and fatigue while investigating self-reported memory failures in cancer patients.

Despites the importance of PM, there have been, to our knowledge, only few studies evaluating PM complaints or PM functioning in patients diagnosed with an intracerebral tumor (such as Diffuse Low-Grade Glioma- DLGG- or glioblastome- GB) or extra-cerebral tumor (such as breast cancer - BC). Therefore, the investigators thought it would be useful, as a first step, to conduct a study to explore and to manage the PM and RM subjective complaints in cancer patients compared to another chronic disease, such as HIV. In fine, these data will help to identify a new target for psychological management focused on either psychopathological or neuropsychological rehabilitation

DETAILED DESCRIPTION:
Primary objective :

This study will aim at determining the nature of subjective memory complaints (i.e., prospective or retrospective memory) in cancer patients with intra- cerebral tumors (Glioblastomas and Diffuse Low Grade Gliomas) and extra cerebral tumors (Breast cancer) compared with controls.

The protocol administration will take about 20 minutes. It will be conducted by an experienced clinical neuropsychologist or clinical oncologist in each center during standard care. According to the results on the questionnaires and test, patients will be addressed and managed by a neuropsychologist, a clinical psychologist, psychiatrist or a speech therapist.

ELIGIBILITY:
Inclusion Criteria:

All the participants must fulfill all the following criteria to be eligible for study entry:

* Be aged of 18 to 80 years old
* Have a ECOG Performance Status ≤ 2 or a Karnofsky index ≥ 50 %
* Have a satisfactory level of French
* Have signed the informed consent

Also, for the DLGG group, the patients must:

* Have a histologically-proven diagnosis of DLGG (i.e., WHO grade II glioma)
* Receive or have received a first oncological treatment after surgery (chemotherapy, radiation therapy…)

Also, for the GB group, the patients must:

- Have a histologically-proven diagnosis of GB (i.e., WHO grade IV glioma).

Also, for the breast cancer group, the patients must:

- Have a histologically-proven diagnosis of breast cancer diagnosed < 2 years.

Exclusion Criteria:

Participants presenting with any of the following exclusion criteria will not be included in the study:

* Patients with brain metastases
* Patients under tutorship or curatorship or protective measures
* Patients suffering from sensorial or motor deficits avoiding the tests administration
* Patients with a reported history of psychiatric disease (e.g., mental retardation, psychotic disorders, learning disabilities, attention-deficit/hyperactivity disorder, and bipolar disorder)
* Have reported a substance dependence within the past six months (e.g., cocaine or methamphetamine dependence)
* Pregnant women
* Legal incapacity or physical, psychological social or geographical status interfering with the patient's ability to sign the informed consent or to terminate the study

Also, for the DLGG group, the patients must not:

* Have an anaplastic glioma (i.e., WHO grade III glioma)
* Have a DLGG with radiological or histological signs of anaplastic transformation
* Have a history of HIV
* Have a history of other cancer

Also, for the GB group, the patients must not:

* Patients treated with ≥2 lines of systemic cancer treatment (e.g., patient after the first GB recurrence)
* Have a history of HIV
* Have a history of other cancer

Also, for the breast cancer group, the patients must not:

* Have a metastatic disease
* Have a neoadjuvant therapy
* Have a documented neurological, or substance use disorders.
* Have a history of HIV
* Have a history of other cancer
* Have reported a history of neurological diagnoses (e.g., seizure disorders, closed head injuries with loss of consciousness greater than 15 min).

Also for the control group, the participants must not:

* Have a documented neurological, or substance use disorders
* Have a history of cancer
* Have a history of HIV

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 426 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
the nature of subjective memory complaints | 12 months
  scores from 8 to 40 of QMRP questionnaire

SECONDARY OUTCOMES:
the significant psychopathological correlates of the subjective PM and RM complaints | 12 months
  Scores on the Hospital Anxiety Depression Scale from 0-21
the significant correlates between the subjective PM and RM complaints and the subjective fatigues | 12 months
  Scores on the Multidimensional Fatigue Inventory-20
the significant correlates between the subjective PM and RM complaints | 12 months
  Scores (from 0 to 30) on the Montreal Cognitive Assessment
the effect of disease on the subjective PM and RM complaints | 12 months
  comparison of clinical event between each group
the effect of cancer on the subjective PM and RM complaints | 12 months
  questionnaire : frontal assessment battery compared between each groups
the significant correlates between the subjective PM and RM complaints | 12 months
  questionnaire : frontal assessment battery score 0-18

CONTACTS AND LOCATIONS:
Overall Officials: Guerdoux Estelle, MD, Study Chair — ICM Co. Ltd.
Locations (6):
- France (6):
  - Icm Val D'Aurelle, Montpellier, Herault
  - CHU D'amiens, Amiens, Nord
  - UFR de Psychologie Université de Lille, Villeneuve-d'Ascq, NORD
  - Hôpital d'Instruction des Armées, Clamart
  - Hopital saint Louis, Paris
  - CHU Lyon, Saint-Genis-Laval

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients The conditions for data transfer of all or part of the study database are decided by the study sponsor and are the subject of a written contract.

REFERENCES:
- [Background] Bedard M, Verma S, Collins B, Song X, Paquet L. Prospective memory impairment in chemotherapy-exposed early breast cancer survivors: Preliminary evidence from a clinical test. J Psychosoc Oncol. 2016 Jul-Aug;34(4):291-304. doi: 10.1080/07347332.2016.1181133. Epub 2016 Apr 28. PMID 27123566
- [Background] Boone M, Roussel M, Chauffert B, Le Gars D, Godefroy O. Prevalence and profile of cognitive impairment in adult glioma: a sensitivity analysis. J Neurooncol. 2016 Aug;129(1):123-30. doi: 10.1007/s11060-016-2152-7. Epub 2016 May 30. PMID 27241133
- [Background] Brem S, Meyers CA, Palmer G, Booth-Jones M, Jain S, Ewend MG. Preservation of neurocognitive function and local control of 1 to 3 brain metastases treated with surgery and carmustine wafers. Cancer. 2013 Nov 1;119(21):3830-8. doi: 10.1002/cncr.28307. Epub 2013 Aug 23. PMID 24037801
- [Background] Cheng H, Yang Z, Dong B, Chen C, Zhang M, Huang Z, Chen Z, Wang K. Chemotherapy-induced prospective memory impairment in patients with breast cancer. Psychooncology. 2013 Oct;22(10):2391-5. doi: 10.1002/pon.3291. Epub 2013 May 15. PMID 23674402
- [Background] Crawford JR, Henry JD, Ward AL, Blake J. The Prospective and Retrospective Memory Questionnaire (PRMQ): latent structure, normative data and discrepancy analysis for proxy-ratings. Br J Clin Psychol. 2006 Mar;45(Pt 1):83-104. doi: 10.1348/014466505X28748. PMID 16480568
- [Background] de Frias CM, Dixon RA, Backman L. Use of memory compensation strategies is related to psychosocial and health indicators. J Gerontol B Psychol Sci Soc Sci. 2003 Jan;58(1):P12-22. doi: 10.1093/geronb/58.1.p12. PMID 12496297
- [Background] Dieckmann P, Reddersen S, Wehner T, Rall M. Prospective memory failures as an unexplored threat to patient safety: results from a pilot study using patient simulators to investigate the missed execution of intentions. Ergonomics. 2006 Apr 15-May 15;49(5-6):526-43. doi: 10.1080/00140130600568782. PMID 16717009
- [Background] Dubois B, Slachevsky A, Litvan I, Pillon B. The FAB: a Frontal Assessment Battery at bedside. Neurology. 2000 Dec 12;55(11):1621-6. doi: 10.1212/wnl.55.11.1621. PMID 11113214
- [Background] Fleming J, Ownsworth T, Doig E, Hutton L, Griffin J, Kendall M, Shum DH. The efficacy of prospective memory rehabilitation plus metacognitive skills training for adults with traumatic brain injury: study protocol for a randomized controlled trial. Trials. 2017 Jan 5;18(1):3. doi: 10.1186/s13063-016-1758-6. PMID 28057075
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Gentile S, Delaroziere JC, Favre F, Sambuc R, San Marco JL. Validation of the French 'multidimensional fatigue inventory' (MFI 20). Eur J Cancer Care (Engl). 2003 Mar;12(1):58-64. doi: 10.1046/j.1365-2354.2003.00295.x. PMID 12641557
- [Background] Gonneaud J, Kalpouzos G, Bon L, Viader F, Eustache F, Desgranges B. Distinct and shared cognitive functions mediate event- and time-based prospective memory impairment in normal ageing. Memory. 2011 May;19(4):360-77. doi: 10.1080/09658211.2011.570765. PMID 21678154
- [Background] Guerdoux E, Dressaire D, Martin S, Adam S, Brouillet D. Habit and recollection in healthy aging, mild cognitive impairment, and Alzheimer's disease. Neuropsychology. 2012 Jul;26(4):517-33. doi: 10.1037/a0028718. Epub 2012 May 28. PMID 22642394
- [Background] Guerdoux E, Martin S, Dressaire D, Adam S, Brouillet D. [Memory controlled processes between the young and old: the birth of cognitive complaint?]. Can J Aging. 2009 Mar;28(1):5-20. doi: 10.1017/S0714980809090023. French. PMID 19860963
- [Background] Herrmann C. International experiences with the Hospital Anxiety and Depression Scale--a review of validation data and clinical results. J Psychosom Res. 1997 Jan;42(1):17-41. doi: 10.1016/s0022-3999(96)00216-4. PMID 9055211
- [Background] Kim HJ, Barsevick AM, Fang CY, Miaskowski C. Common biological pathways underlying the psychoneurological symptom cluster in cancer patients. Cancer Nurs. 2012 Nov-Dec;35(6):E1-E20. doi: 10.1097/NCC.0b013e318233a811. PMID 22228391
- [Background] Kliegel M, Altgassen M, Hering A, Rose NS. A process-model based approach to prospective memory impairment in Parkinson's disease. Neuropsychologia. 2011 Jul;49(8):2166-77. doi: 10.1016/j.neuropsychologia.2011.01.024. Epub 2011 Jan 19. PMID 21255592
- [Background] Kliegel M, Martin M, McDaniel MA, Einstein GO. Varying the importance of a prospective memory task: differential effects across time- and event-based prospective memory. Memory. 2001 Jan;9(1):1-11. doi: 10.1080/09658210042000003. PMID 11315657
- [Background] Kvavilashvili L, Kornbrot DE, Mash V, Cockburn J, Milne A. Differential effects of age on prospective and retrospective memory tasks in young, young-old, and old-old adults. Memory. 2009 Feb;17(2):180-96. doi: 10.1080/09658210802194366. PMID 18608976
- [Background] Lange M, Joly F. How to Identify and Manage Cognitive Dysfunction After Breast Cancer Treatment. J Oncol Pract. 2017 Dec;13(12):784-790. doi: 10.1200/JOP.2017.026286. PMID 29232539
- [Background] Martin S, Mazzocco C, Maury P, Grosselin A, Van der Elst W, Dixon RA, Brouillet D. Compensating for memory losses throughout aging: validation and normalization of the memory compensation questionnaire (MCQ) for non-clinical French populations. Arch Gerontol Geriatr. 2015 Jan-Feb;60(1):28-38. doi: 10.1016/j.archger.2014.10.013. Epub 2014 Oct 22. PMID 25459917
- [Background] Meyers CA, Wefel JS. The use of the mini-mental state examination to assess cognitive functioning in cancer trials: no ifs, ands, buts, or sensitivity. J Clin Oncol. 2003 Oct 1;21(19):3557-8. doi: 10.1200/JCO.2003.07.080. Epub 2003 Aug 11. No abstract available. PMID 12913103
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Paquet L, Collins B, Song X, Chinneck A, Bedard M, Verma S. A pilot study of prospective memory functioning in early breast cancer survivors. Breast. 2013 Aug;22(4):455-61. doi: 10.1016/j.breast.2013.04.002. Epub 2013 May 4. PMID 23648279
- [Background] Paquet L, Verma S, Collins B, Chinneck A, Bedard M, Song X. Testing a novel account of the dissociation between self-reported memory problems and memory performance in chemotherapy-treated breast cancer survivors. Psychooncology. 2018 Jan;27(1):171-177. doi: 10.1002/pon.4389. Epub 2017 Feb 10. PMID 28129471
- [Background] Woods SP, Moran LM, Dawson MS, Carey CL, Grant I; HIV Neurobehavioral Research Center (HNRC) Group. Psychometric characteristics of the memory for intentions screening test. Clin Neuropsychol. 2008 Sep;22(5):864-78. doi: 10.1080/13854040701595999. PMID 18756389
- [Background] Razavi D, Delvaux N, Farvacques C, Robaye E. Screening for adjustment disorders and major depressive disorders in cancer in-patients. Br J Psychiatry. 1990 Jan;156:79-83. doi: 10.1192/bjp.156.1.79. PMID 2297623
- [Background] Scullin MK, McDaniel MA, Shelton JT. The Dynamic Multiprocess Framework: evidence from prospective memory with contextual variability. Cogn Psychol. 2013 Aug-Sep;67(1-2):55-71. doi: 10.1016/j.cogpsych.2013.07.001. Epub 2013 Aug 3. PMID 23916951
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775
- [Background] Smith G, Della Sala S, Logie RH, Maylor EA. Prospective and retrospective memory in normal ageing and dementia: a questionnaire study. Memory. 2000 Sep;8(5):311-21. doi: 10.1080/09658210050117735. PMID 11045239
- [Background] Smith T, Gildeh N, Holmes C. The Montreal Cognitive Assessment: validity and utility in a memory clinic setting. Can J Psychiatry. 2007 May;52(5):329-32. doi: 10.1177/070674370705200508. PMID 17542384
- [Background] Woods SP, Carey CL, Moran LM, Dawson MS, Letendre SL, Grant I; HIV Neurobehavioral Research Center (HNRC) Group. Frequency and predictors of self-reported prospective memory complaints in individuals infected with HIV. Arch Clin Neuropsychol. 2007 Feb;22(2):187-95. doi: 10.1016/j.acn.2006.12.006. Epub 2007 Feb 6. PMID 17289343
- [Background] Zeintl M, Kliegel M, Rast P, Zimprich D. Prospective memory complaints can be predicted by prospective memory performance in older adults. Dement Geriatr Cogn Disord. 2006;22(3):209-15. doi: 10.1159/000094915. Epub 2006 Aug 7. PMID 16899998
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820